CLINICAL TRIAL: NCT07391267
Title: Pathogenesis of Chronic Kidney Disease Associated With Metabolic Dysfunction- Associated Fatty Liver Disease (MAFLD) and Treatment Response of Oral Semaglutide - a Randomized Controlled Trial.
Brief Title: Pathogenesis of Chronic Kidney Disease Associated With Metabolic Dysfunction- Associated Fatty Liver Disease (MAFLD) and Treatment Response of Oral Semaglutide.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-CKD-01
Record Dates: First submitted 2025-12-15; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Diseases; MAFLD
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Patient and Investigator
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Medical Treatment (SMT) (Active Comparator): Control arm : Participants in this arm will receive Placebo with Standard Medical Treatment (SMT).
  Interventions: Other: Placebo; Other: Standard medical treatment
- Semaglutide with Standard Medical Treatment (Experimental): Semaglutide with Standard Medical Treatment: Participants in this arm will receive Standard medical treatment and oral semaglutide starting from 3mg dose daily that gradually increases upto 14mg dose daily for 6 months.
  Interventions: Drug: Semaglutide Oral Tablet; Other: Standard medical treatment

INTERVENTIONS:
Drug: Semaglutide Oral Tablet — GLP1-R agonists GLP1-R agonists (GLP1-RAs) are novel potent antidiabetic agents with proven efficacy in reducing major adverse cardiovascular events. Besides their glucose-lowering action, their beneficial hepatic effects may be related to the influence on the AMPK/mTOR pathway. Semaglutide was associated with significant decreases in body weight, alanine aminotransferase, liver steatosis, and stiffness.GLP1-RAs may also improve histologic features on NAFLD, such as liver fat deposition, steatohepatitis, and fibrosis. GLP1-RAs have shown benefits in preventing the development or halting the progression of CKD. It also promotes antioxidative and anti-inflammatory actions may be among the determining factors in this renoprotective effect, together with weight loss, blood pressure, and glucose-lowering.
  Arms: Semaglutide with Standard Medical Treatment
Other: Placebo — Placebo will be given in the same manner.
  Arms: Standard Medical Treatment (SMT)
Other: Standard medical treatment — Standard medical treatment-
  1. Lifestyle first - weight loss , caloric restriction, increased aerobic + resistance exercise, treat obesity and metabolic syndrome.
  2. Optimize blood-pressure control and use RAAS blockade when indicated (ACE inhibitor or ARB) to reduce albuminuria and slow CKD progression .
  3. Treat dysglycaemia and favour drug classes with kidney + liver benefit when appropriate
     * SGLT2 inhibitors (dapagliflozin, empagliflozin, canagliflozin) - recommended for people with T2D + CKD
     * GLP-1 receptor agonists (e.g., semaglutide)
  4. Lipid management / statins - treat according to CV risk
  5. Consider established liver-directed agents when appropriate
  6. Pioglitazone (thiazolidinedione) and vitamin-E
  7. Standard CKD supportive care - salt and fluid management, correction of metabolic acidosis, anaemia and mineral bone abnormalities as per CKD stage; immunize and address CV risk factors aggressively
  8. Avoid hepatotoxic drugs / review medications

SUMMARY:
This project aims to investigate how Chronic Kidney Disease (CKD) develops and progresses in patients who also have Non-Alcoholic Fatty Liver Disease (NAFLD) and to evaluate whether oral semaglutide (a GLP-1 receptor agonist) can slow or prevent this progression.

NAFLD and CKD frequently coexist due to shared mechanisms such as insulin resistance, inflammation, oxidative stress, dyslipidemia, and metabolic syndrome. Because of these overlapping pathways, a single therapy targeting both organs may offer major benefits.

Semaglutide is known to reduce liver fat, improve inflammation and fibrosis, promote weight loss, and provide renal protection. This project will test whether adding oral semaglutide to standard care leads to better kidney and liver outcomes than standard care alone.

The study is designed as a randomised controlled trial conducted at ILBS, enrolling adults having NAFLD with CKD (with specific eGFR and albuminuria criteria). Participants will be followed for 2 years, with regular assessment of kidney function (eGFR, ACR), liver health (FibroScan, ALT/AST), metabolic parameters, and cardiovascular outcomes.

A parallel animal study in mice with diet-induced fatty liver disease will validate mechanistic findings through liver and kidney histology, gene expression, metabolic tests, and biochemical markers after semaglutide treatment.

Expected outcome: To demonstrate that semaglutide slows CKD progression and improves NAFLD, supporting its use as a therapeutic option for patients with coexisting both conditions.

DETAILED DESCRIPTION:
NAFLD and metabolic syndrome have emerged as significant health concerns globally, with substantial implications for kidney health.The interplay between NAFLD, metabolic syndrome, and CKD necessitates a comprehensive understanding of the underlying mechanisms and shared pathogenic pathways. Their shared risk factors, molecular mechanisms, and genetic predisposition represent the basis for this relationship.

Accordingly, treatment approaches with combined efficacy in NAFLD and chronic renal impairment are expected to positively impact the natural history of this deleterious interaction.

GLP1-R agonists GLP1-R agonists (GLP1-RAs) are novel potent antidiabetic agents with proven efficacy in reducing major adverse cardiovascular events. Besides their glucose-lowering action, their beneficial hepatic effects may be related to the influence on the AMPK/mTOR pathway. Semaglutide was associated with significant decreases in body weight, alanine aminotransferase, liver steatosis, and stiffness.GLP1-RAs may also improve histologic features on NAFLD, such as liver fat deposition, steatohepatitis, and fibrosis. GLP1-RAs have shown benefits in preventing the development or halting the progression of CKD. It also promotes antioxidative and anti-inflammatory actions may be among the determining factors in this renoprotective effect, together with weight loss, blood pressure, and glucose-lowering.

Primary objective-To measure the progression of CKD and NAFLD in Semaglutide treated group versus non treated group.

Secondary objectives-1.To conduct animal model studies to confirm the primary objective by performing the liver and renal histology.

Study Population-All patients diagnosed to have NAFLD with or without DM Type2 with CKD(GFR<60 ML/MIN AND ALBUMINURIA (>330 MG/MMOL)will be included in the study.

STUDY PLAN Type of study-Randomised Control Trial(RCT) Study period-3 years Intervention-adding oral semaglutide once a day (starting from 3mg to 14 mg ).we will start from 3mg once a day and go upto 14 mg once a day . Control arm-patients receiving standard of care.

Statistical analysis: Categorical values were reported as numbers, frequencies and percentages. Continuous data was reported as median and interquartile range (IQR) or mean with standard deviation. Chi square/Chi square with yate's correction/Fisher test was used for comparing categorical values depending on the sample size. For comparing continuous data, unpaired t-test or Mann Whitney was used as appropriate16 was used for statistical analysis. A p-value of below 0.05 was adapted as a value of statistical significance for the purpose of this study.Intension to treat and per protocol analysis will be done and any adverse event will be reported.

ANIMAL MODEL Male C57BL/6J mice (6 weeks old) are selected for the study Mice will be induced to liver disease by feeding a rodent diet with 58 Kcal% fat and sucrose (D12331- Research diets) for 20- 32 weeks and Mice on a standard chow diet will be included as controls. 6-week-old mice will be fed with 50% supplementation of a High-fat diet with standard chow diet for acclimatization for period of two weeks. Post which a complete high fat diet will be administered.

To reflect the disease state at the start of treatment, animals will be sacrificed from both groups. Histology for liver and kidney will be performed at dose start (baseline group), other endpoints and biochemical parameters will also be analyzed at this point.

Oral animal equivalent dose will be calculated using known human dose of Semaglutide. Oral semaglutide pills will be crushed into powder form and resuspended in distilled water for oral gavage. Semaglutide or vehicle (Distilled water/ Normal saline) will be administered orally daily for 8-12 weeks, while body weight, food and water consumption will be monitored daily. Weekly Insulin tolerance test and glucose tolerance test will be performed from the start of 20th weeks to analyze insulin resistance and hyperglycemia in mice model.

At study termination, blood sampled via retro-orbital will be collected for analysis of liver enzymes, plasma lipids (ALT, AST, TG and TC), serum urea, creatinine, and blood urea nitrogen. Urine will be collected to measure Albumin and creatinine using commercially available ELISA kits. Collected plasma samples will be used to measure levels of Adiponectin, leptin, resistin and ghrelin using commercially available ELISA kits. Animals will be euthanized using ketamine and xylazine cocktail, and liver and renal tissues will be collected weighed and subjected to histology, gene expression and other biochemical parameters for further study and inference.

These expected deliverable aim to demonstrate the efficacy of Semaglutide in slowing the progression of CKD and NAFLD, validated through both clinical and preclinical studies, thereby supporting its potential use as a therapeutic option for these conditions.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age above or equal to 18 years at the time of signing informed consent. 2.Diagnosed with type 2 diabetes mellitus 3.HbA1c less than or equal to 10% (less than or equal to 86 mmol/mol) 4.Renal impairment defined either by:
* serum creatinine-based eGFR greater than or equal to 50 and less than or equal to 75 mL/min/1.73 m^2 (CKD-EPI) and UACR greater than 300 and less than 5000 mg/g or
* serum creatinine-based eGFR greater than or equal to 25 and less than 50 mL/min/1.73 m^2 (CKD-EPI) and UACR greater than 100 and less than 5000 mg/g 5.Treatment with maximum labelled or tolerated dose of a reninangiotensin-aldosterone system (RAAS) blocking agent including an angiotensin converting enzyme (ACE) inhibitor or an angiotensin II receptor blocker (ARB), unless such treatment is contraindicated or not tolerated. Treatment dose must be stable for at least 4 weeks prior to the date of the laboratory assessments used for determination of the inclusion criteria for renal impairment and kept stable until screening.

Exclusion Criteria:

1. Documented causes of chronic liver disease other than non-alcoholic fatty liver disease (NAFLD)
2. Positive HBsAg, positive anti-HIV, positive HCV RNA at screening (V2A) or any known presence of HCV RNA or HBsAg within 2 years of screening (V2A).
3. Presence or history of ascites, variceal bleeding, hepatic encephalopathy, spontaneous bacterial peritonitis or liver transplantation at randomisation.
4. Known or suspected excessive consumption of alcohol (greater than 20 g/day for women or greater than 30 g/day for men) or alcohol dependence (assessed by the Alcohol Use Disorders Identification Test (AUDIT questionnaire)).
5. Treatment with vitamin E (at doses greater than or equal to 800 IU/day) or pioglitazone or medications approved for treatment of NASH which has not been at a stable dose in the period from 90 days prior to the screening visit (V2A). In addition, for subjects with historical liver biopsies taken more than 90 days prior to screening, treatment should be at a stable dose from time of biopsy until screening.
6. Treatment with GLP-1 RAs in the period from 90 days prior to the screening visit (V2A). In addition, for subjects with historical liver biopsies taken more than 90 days prior to screening, any treatment with GLP-1 RAs from time of biopsy until screening (V2A).
7. Treatment with glucose-lowering agent(s) (other than GLP-1 RAs), lipid-lowering medication or weight loss medication not stable in the opinion of the investigator in the period from 90 days prior to the screening visit (V2A). In addition, for subjects with historical liver biopsies taken more than 90 days prior to screening, treatment should be at a stable dose in the opinion of the investigator from time of biopsy until screening.
8. Congenital or hereditary kidney diseases including polycystic kidney disease, autoimmune kidney diseases including glomerulonephritis or congenital urinary tract malformations
9. Myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within 60 days prior to the day of screening.
10. Presently classified as being in New York Heart Association (NYHA) Class IV heart failure
11. Planned coronary, carotid or peripheral artery revascularisation
12. Current (or within 90 days) chronic or intermittent haemodialysis or peritoneal dialysis 13 Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupildilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of a composite primary outcome event defined as persistent eGFR decline of greater than or equal to 50 percentage from trial start, reaching ESRD, death from kidney disease or death from cardiovascular disease. | 3 months, 6 months, 12 months,18 months and 24 months

SECONDARY OUTCOMES:
Annual rate of change in eGFR (chronic kidney disease - epidemiology collaboration (CKD-EPI)) | 3 months, 6 months, 12 months,18 months and 24 months
ime to first occurrence of a composite cardiovascular major adverse cardiovascular event (MACE) endpoint consisting of: Non-fatal myocardial infarction, non-fatal stroke, and cardiovascular (CV) death | 3 months, 6 months, 12 months,18 months and 24 months
Time to occurrence of all-cause death | 3 months, 6 months, 12 months,18 months and 24 months
Change in eGFR and proteinuria. | 3 months, 6 months, 12 months,18 months and 24 months
Annual rate of change in eGFR (CKD-EPI) (chronic eGFR slope) | 3 months, 6 months, 12 months,18 months and 24 months
Change in eGFR (CKD-EPI) and cystatin C | 3 months, 6 months, 12 months,18 months and 24 months
Change in albumin creatinine ratio(ACR) | 3 months, 6 months, 12 months,18 months and 24 months
Change in bodyweight | 3 months, 6 months, 12 months,18 months and 24 months
Change in HBA1c | 3 months, 6 months, 12 months,18 months and 24 months
Change in Systolic and diastolic BP | 3 months, 6 months, 12 months,18 months and 24 months
Number of hypoglycemic episodes | 3 months, 6 months, 12 months,18 months and 24 months
Changes in the liver histology in the animal model as assessed by Alpha-SMA, Col-1. | 4,8,16,24 weeks
Changes in the liver histology in the animal model as assessed by SGOT/SGPT. | 4,8,16,24 weeks
Changes in the renal histology in the animal model as assessed by UPCR,GFR,Creatinine clearance. | 4,8,16,24 weeks
Changes in the renal histology in the animal model as assessed by FITC-Sinistrin Clearance,cystatin-C. | 4,8,16,24 weeks
Resolution of steatohepatitis and improvement in liver fibrosis (Yes/No) | 3 months, 6 months, 12 months,18 months and 24 months
Changes in liver stiffness values assessed by transient elastography (FibroScan®) | 3 months, 6 months, 12 months,18 months and 24 months
Change in ELF (Enhanced Liver Fibrosis) score | 3 months, 6 months, 12 months,18 months and 24 months
Change in ALT/AST | 3 months, 6 months, 12 months,18 months and 24 months
Change in CAP (Controlled Attenuation Parameter) values assessed by transient elastography (FibroScan) | 3 months, 6 months, 12 months,18 months and 24 months
Change in FAST (FibroScan-AST) score | 3 months, 6 months, 12 months,18 months and 24 months
Change in inflammation assessed by hsCRP (High Sensitive C-Reactive Protein) | 3 months, 6 months, 12 months,18 months and 24 months
Change in triglyceride/LDL | 3 months, 6 months, 12 months,18 months and 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India